CLINICAL TRIAL: NCT01333462
Title: A Phase 1 Randomized, Single-Blind, Controlled, Safety, Tolerability and Immunogenicity Study of Intranasal NB-1008 (Fluzone® + 60%W805EC) in Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity Study of Inactivated Nasal Influenza Vaccine NB-1008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Jakub Simon, MD, MS/ Director, Clinical Vaccine Development, NanoBio Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NB-1008-001
Record Dates: First submitted 2011-04-05; First posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (12):
- Phosphate Buffered Saline (PBS) IN (Placebo Comparator)
  Interventions: Other: Control
- Fluzone 4 mcg HA IN (Active Comparator)
  Interventions: Other: Control
- Fluzone 15 mcg HA IM (Active Comparator)
  Interventions: Other: Control
- NB-1008 4 mcg HA 5% W805EC (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 4 mcg HA 10% W805EC (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 4 mcg HA 15% W805EC (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 4 mcg HA 20% W805EC (Experimental)
  Interventions: Biological: NB-1008
- Fluzone 10 mcg HA IN (Active Comparator)
  Interventions: Other: Control
- NB-1008 10 mcg HA 5% W805EC (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 10 mcg HA 10% W805EC (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 10 mcg HA 15% W805EC (Experimental)
  Interventions: Biological: NB-1008
- NB-1008 10 mcg HA 20% W805EC (Experimental)
  Interventions: Biological: NB-1008

INTERVENTIONS:
Biological: NB-1008 — NB-1008 is composed of Fluzone containing 4 micrograms (mcg) or 10 micrograms of strain-specific hemagglutinin (HA) and 5%, 10%, 15%, or 20% W805EC adjuvant.
  Arms: NB-1008 10 mcg HA 10% W805EC; NB-1008 10 mcg HA 15% W805EC; NB-1008 10 mcg HA 20% W805EC; NB-1008 10 mcg HA 5% W805EC; NB-1008 4 mcg HA 10% W805EC; NB-1008 4 mcg HA 15% W805EC; NB-1008 4 mcg HA 20% W805EC; NB-1008 4 mcg HA 5% W805EC
Other: Control — The controls include PBS placebo control as well as Fluzone IN and IM active controls.
  Arms: Fluzone 10 mcg HA IN; Fluzone 15 mcg HA IM; Fluzone 4 mcg HA IN; Phosphate Buffered Saline (PBS) IN

SUMMARY:
The purpose of this study is to test the safety and immune response of a new intranasal vaccine against influenza, called NB-1008. The vaccine is composed of a licensed vaccine that is normally given as an injection, called Fluzone, and an adjuvant (additive that helps a vaccine work better), called W805EC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Are 18-49 years of age, inclusive.
3. If female, must be non-pregnant as confirmed by a negative serum pregnancy test conducted at screening and a negative urine pregnancy test conducted at the site within 24 hours preceding receipt of vaccine.
4. Females who are not surgically sterile or at least one year post-menopausal agree to use oral, implantable, transdermal or injectable contraceptive or another reliable form of contraception approved by the Investigator for a minimum of 30 days prior to vaccination and for 3 months following vaccination.
5. Healthy, as determined by medical history, physical examination, vital signs, and clinical laboratory examinations.
6. Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
7. Has given written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of significant acute or chronic, uncontrolled medical or psychiatric illness (institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months). Subjects with a history of chronic cough, frequent sinus infections, sinusitis, allergic rhinitis, nasal polyps or obstruction, including deviated septum significant enough to obstruct the nasal openings are to be excluded. Subjects with seasonal rhinitis may be included if their 'season' does not occur within 3 months of the vaccination date and they are not currently receiving intranasal steroids.
2. Receipt of the 2008-2009 influenza vaccine.
3. Positive serology for HIV-1 or HIV-2, or HCV antibodies.
4. Platelet count <150,000/mm3.
5. Positive urine drug screen.
6. History of aspiration, dysphagia, swallowing disorders, stroke or other neurologic conditions that may predispose the subject to aspiration of test articles into the respiratory tract.
7. History of Bell's palsy.
8. Cancer or treatment for cancer, within 3 years. Subjects with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Basal cell carcinoma (BCC) or (SCC) are allowed, unless present on or near the nose.
9. Impaired immune responsiveness, regardless of cause, including diabetes mellitus.
10. Presently receiving or history of receiving any medications or treatments that affects the immune system such as immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months.
11. Chronic use of inhaled or intranasal sprays including decongestants and corticosteroids.
12. Presently a smoker or tobacco user or have a history of smoking or tobacco use within the past year prior to screening.
13. Receipt or planned administration of a nonstudy vaccine within 30 days before the study, including licensed influenza vaccines and prior to the Day 60 telephone contact. Immunization on an emergency basis with Tetanus Toxoids Adsorbed for adult use (Td or Tdap) up to 8 days before or at least 8 days after a dose of study vaccine will be allowed. Administration of study vaccine can be delayed if a nonstudy vaccine has been administered and will be given as soon as acceptable, as described above.
14. Known allergy to any vaccine component, including eggs, egg products, or thimerosal.
15. History of allergic and/or anaphylactic type reaction to injected vaccines or to any of the components of NB-1008 [soybean oil, dehydrated alcohol (anhydrous ethanol), polysorbate (Tween 80) and cetylpyridinium chloride (CPC)].
16. History of drug or chemical abuse in the year before the study.
17. Receipt of any investigational product or nonregistered drug within the 30 days before study entry or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing 6 month period.
18. Use of nasally administered prescription or over-the-counter (OTC) medications within 7 days before vaccination
19. Receipt of blood or blood products 8 weeks before study entry or planned administration prior to the Day 60 telephone contact.
20. Donation of blood or blood products within 8 weeks before study entry or at any time up to the Day 28 clinic visit.
21. Acute disease within a week prior to vaccination, defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination) with or without fever. For subjects with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade febrile illness, the subject can be re-screened once they have complexly recovered.
22. Any condition that, in the opinion of the investigator, might interfere with study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 365 Days
  Adverse events (AE) collected through Day 28 and Serious Adverse Events (SAE) collected through Day 365.

SECONDARY OUTCOMES:
Serum hemagglutination-inhibition (HAI) Geometric Mean Titer (GMT) and proportion of Volunteers with >=4 fold increase in titer as well as proportion of volunteers with titer >= protective level of 40 | Day 28 and Day 60
  HAI antibody titers to H1N1, H3N2, and B influenza strains contained in the vaccine.
Nasal wash anti-Fluzone IgA Geometric Mean Titer (GMT) and proportion of volunteers with >=4 fold increase in GMT anti-Fluuzone IgA titer | Day 28 and Day 60
  Nasal Wash IgA to Fluzone.

CONTACTS AND LOCATIONS:
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States